CLINICAL TRIAL: NCT00850369
Title: A Pilot Study of the Effects of Chronic Red Blood Cell Transfusion in Sickle Cell Disease On Pulmonary Hypertension in Patients With Sickle Cell Disease
Brief Title: A Pilot Study of Chronic Red Blood Cell Transfusion in Sickle Cell Disease-Associated Pulmonary Hypertension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual onto the study
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01-HL79915-1; HL799151; R01HL079915 (NIH)
Record Dates: First submitted 2009-02-22; First posted 2009-02-25 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Hypertension; Sickle Cell Disease
Keywords: Pulmonary hypertension; Sickle cell disease
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All subjects wil receive monthly RBC transfusions for 6 months
  Interventions: Other: RBC transfusion

INTERVENTIONS:
Other: RBC transfusion — Study subjects will receive monthly transfusions with 2 units of red blood cells

SUMMARY:
Pulmonary hypertension, a complication associated with an increased risk of death, is common in patients with sickle cell disease. Despite its frequency, there remains no standard treatment for this complication in patients with sickle cell disease.

In this small study, the investigators will evaluate the effect of monthly transfusion of red blood cells to patients with sickle cell disease-associated pulmonary hypertension. The investigators speculate that by increasing the hemoglobin level and decreasing the amount of sickle red blood cells, these patients would experience improvements in their PHT.

DETAILED DESCRIPTION:
As patients with sickle cell disease (SCD) age, recurrent vaso-occlusive episodes lead to progressive end-organ damage. Pulmonary hypertension (PHT) represents an example of such end-organ damage. Pulmonary hypertension, a common complication in patients with sickle cell disease (SCD), results in a shortened survival. The high mortality reported in SCD patients with PHT appears to occur particularly in those patients with moderate and severe elevations in their pulmonary artery pressure. The overall objective of this proposal is to evaluate the effect of chronic red blood cell transfusion on PHT in SCD. We hypothesize that by increasing the hemoglobin concentration and decreasing the amount of HbS, these patients would experience improvements in their PHT.

Thus, the specific aim of this clinical trial is to evaluate the effects of RBC transfusion on pulmonary hypertension in SCD, as well as the effect of chronic RBC transfusion on plasma markers of thrombin generation, platelet activation, and nitric oxide metabolites.

Study subjects will be transfused monthly for 6 months to investigate the safety and efficacy of RBC transfusion in SCD patients with PHT. All packed red blood cells will have extended antigen matching for C, D, E and Kell to minimize the risk of alloimmunization. Subjects will receive other routine treatments for SCD. Specific outcome variables will be evaluated at 1 month, 3 months, and 6 months. All study subjects will receive simple transfusion of packed red blood cell to achieve a post-transfusion hemoglobin (Hb) not greater than 10 g/dL. For those subjects who may have baseline hemoglobins in whom a post transfusion Hb would exceed 10 g/dL, they will require a limited exchange transfusion, i.e. phlebotomy of 1 unit of blood, followed by transfusion of 2 units of packed RBC. All study subjects will return for assessment of safety and/or efficacy measures every two weeks for the first month, and subsequently every four weeks till the completion of the study. Study subjects who experience a documented worsening of their disease (decreased SaO2, worsening 6-minute walk) on at least two consecutive follow up visits will be taken off the study. At the end of the study, subjects will have the option of continuing on chronic RBC transfusion.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of sickle cell anemia (HbSS) and HbSbeta0 thalassemia;
2. male and female subjects between 18 and 65 years;
3. documented PHT, but with pulmonary artery systolic pressures >/= 45 mmHg (TR jet velocity of >/= 3.0 m/s) on at least 2 separate visits at least 1 month apart;
4. ability to give written informed consent to participate in the study; and
5. in non-crisis steady state at time of enrollment

Exclusion Criteria:

1. treatment with epoprostenol (flolan) or similar prostacyclin analog, bosentan or sildenafil (or similar phosphodiesterase 5 inhibitor)
2. on chronic anticoagulation
3. RBC transfusion in previous 90 days;
4. use of hydroxyurea
5. multiple red cell alloantibodies that will make transfusion unsafe;
6. baseline ferritin level > 1000 mg/dL
7. pregnancy, and/or any condition which in the opinion of investigator might make the subject unsuitable for the study;
8. patients with WHO functional class IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery systolic pressure (mm Hg) | 2 years
Pulmonary vascular resistance (dyne.s.cm-5) | 2 years

SECONDARY OUTCOMES:
Six-minute walk | 2 years
Markers of thrombin generation (TAT complexes, F1.2, d-dimers) | 2 years
Markers of platelet activation (soluble CD40 ligand, beta thromboglobulin, platelet factor | 2 years
Nitric oxide metabolites | 2 years
Quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MD, Principal Investigator — University of North Carolina, Chapel Hill